CLINICAL TRIAL: NCT07236567
Title: Evaluation of the Effect of Grape Seed Extract, Glycyrrhizin Compared to Triple Antibiotic Paste as Intra Canal Medication in Revascularization of Necrotic Permanent Immature Teeth in Children: A Randomized Clinical Trial
Brief Title: Revascularization of Young Immature Permenant Teeth Using Different Types of Intra Canal Medication
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Mohamed Khalifa, Doctor of dental medicine, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Revascularization
Record Dates: First submitted 2025-11-15; First posted 2025-11-19 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Traumatic Teeth; Necrotic Teeth
Keywords: Revascularization; Grape seed extract; Glycyrrhizin
MeSH Terms: interventions — Grape Seed Extract; Glycyrrhizic Acid

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group a (Active Comparator): Revascularization with triple antibiotic paste as intracanal medication
  Interventions: Drug: Triple Antibiotic Paste
- Group b (Experimental): Revascularization with grape seed extract as intra canal medication
  Interventions: Drug: Grape Seed Extract
- Group c (Experimental): Revascularization with glycyrrhizin as intracanal medication
  Interventions: Drug: Glycyrrhizin

INTERVENTIONS:
Drug: Grape Seed Extract — Grape seed extract in form of hydrogel with concentration 6.5 % left in canal for one week
  Arms: Group b
Drug: Glycyrrhizin — Glycyrrhizin hydrogel 50 micrograms in 1 milligram left in canal for one week
  Arms: Group c
Drug: Triple Antibiotic Paste — Trple antibiotic paste Left for one week
  Arms: Group a

SUMMARY:
Evaluation of the Effect of Grape Seed Extract, Glycyrrhizin Compared to Triple Antibiotic Paste as Intra Canal Medication in Revascularization of Necrotic Permanent Immature Teeth in Children: A Randomized Clinical Trial

DETAILED DESCRIPTION:
Digital count of e.faecalis before and after application of different type of intra canal medication

ELIGIBILITY:
Inclusion Criteria:

* Healthy children aged from 7-13 years old.
* Patient with necrotic pulp.
* Open apex.

Exclusion Criteria:.

* Teeth with root fractures.
* Presence of root resorptions.
* Presence of periodontal pockets.
* Developmental anomalies.
* Tooth with class III mobility

Ages: 7 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 45 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2027-10-01 (Estimated); Study Completion 2027-11-01 (Estimated)

PRIMARY OUTCOMES:
Digital count of e.faecalis | After One week of mediation application
  Microbiological evaluation The number of E. faecalis will be digitally counted.
Clinical evaluation success will be assessed using following criteria of success according to scoring system Absence of : - Pain, - Soft tissue swelling - soft tissue inflammation - Sinus tract - tenderness to percussion - tooth mobility | After one week of mediation application
  Clincal success will be assessed using following criteria of success according to clinical scoring system
  Absence of :
  * Pain,
  * Soft tissue swelling
  * soft tissue inflammation
  * Sinus tract
  * tenderness to percussion
  * tooth mobility. Clinical score Clinical symptom Definition
    1. asymptomatic Pathology: absent Normal functioning Mobility (physiological) ≤1mm
    2. Slight discomfort, short-lived Pathology: questionable Percussion sensitivity Gingival inflammation (due to poor oral hygiene) Mobility (physiological) > 1mm, but <2mm
    3. Minor discomfort, short-lived Pathology: initial changes present Gingival swelling (not due to poor oral hygiene) Mobility > 2mm, but < 3 mm
    4. Major discomfort, long-lived extract immediately Pathology: late changes present Spontaneous pain Gingival swelling (not due to poor oral hygiene) Periodontal pocket formation(exudate) Sinus tract present Mobility ≥ 3mm Premature tooth loss, due to pathology

SECONDARY OUTCOMES:
Radiographic evaluation | After tweleve month
  After tweleve months take periapical radiograph to detection normal lamina dura and increase in root thikness and length. Criteria for success according to radiographic scoring system

CONTACTS AND LOCATIONS:
Locations (1):
- Al-Azhar University faculty of dental medicine, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Evaluation of the Effect of Grape Seed Extract, Glycyrrhizin Compared to Triple Antibiotic Paste as Intra Canal Medication in Revascularization of Necrotic Permanent Immature Teeth in Children: A Randomized Clinical Trial